CLINICAL TRIAL: NCT02257099
Title: Comparison of a Novel Weight Bearing Cone Beam Computed Tomography (CT)Scanner Versus a Conventional CT Scanner for Measuring Patellar Instability
Brief Title: CT Analysis of the Patellofemoral Joint in Patients Having Knee Surgery
Acronym: PF
Status: Completed | Type: Observational
Sponsor: State University of New York at Buffalo (Other)
Collaborators: Carestream Health, Inc. (Industry)
Responsible Party: Principal Investigator, John Marzo, Associate Professor of Clinical Orthopaedics, State University of New York at Buffalo
Other Study IDs: 655951-1
Record Dates: First submitted 2014-09-29; First posted 2014-10-06 (Estimated); Results first posted 2019-10-03 (Actual); Last update posted 2019-10-03 (Actual); Status verified 2019-09

CONDITIONS: Patellar (or Kneecap) Instability and Mal-alignment
MeSH Terms: conditions — Patella Fracture

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No

SUMMARY:
The primary hypothesis is that measures of patellofemoral alignment obtained from the investigational cone beam CT scanner will be reduced, but still correlated to those obtained from the conventional CT scan.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have been diagnosed with acute or chronic patellar malalignment.
* At least 16 years old
* Be willing and able to provide informed consent

Exclusion Criteria:

* Open growth plates
* Previous knee surgery on the affected knee
* Pregnancy (females)
* Fracture of the patellofemoral joint
* Knee ligament injury (other than medial patellofemoral ligament)
* Have greater than Grade II degenerative changes of the patellofemoral joint
* Inability to bear weight on the extremity during the CT scan

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who have been diagnosed with acute or chronic patellar malalignment.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2015-02; Primary Completion 2016-02 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - UBMD Orthopaedics and Sports Medicine, Northtowns office, Amherst, New York
  - UBMD Orthopaedics and Sports Medicine, Southtowns Office, Orchard Park, New York

RESULTS

PARTICIPANT FLOW:
Groups:
- Cases: Case-only, patients with patellar instability and mal-alignment
Period: Overall Study
Arm/Group | Cases
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Patients aged 16 and older diagnosed with patellar instability and mal-alignment
Groups:
- Cases: Case-only study, patients with patellar instability or mal-alignment
Arm/Group | Cases
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4
  Between 18 and 65 years | 16
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.5 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 8
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Congruence Angle CBCT
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: degrees
Groups:
- Conventional CT: conventional CT scan
- CBCT: CBCT scan
Arm/Group | Conventional CT | CBCT
Number analyzed (Participants) | 20 | 20
degrees | 26.7 (18.1) | 3 (30.1)

2. Secondary Outcome: Tilt Angle
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Cases
Number analyzed (Participants) | 20
degrees | 18.2 (11.6)

3. Secondary Outcome: Tibial Tuberosity Trochlear Groove
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Cases
Number analyzed (Participants) | 20
mm | 12.3 (6.3)

ADVERSE EVENTS:
Groups:
- Cases: Case-only study, patients with patellar instability and mal-alignment
Arm/Group | Cases
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No